CLINICAL TRIAL: NCT06068998
Title: Molecular Characterization of Penile Cancers in Developing Countries
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: LACOG 2018
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Penile Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explores penile squamous cell carcinoma (PSCC) in Brazil, a rare cancer associated with factors like poor hygiene and HPV infection, using next-generation sequencing to investigate its genomic profiles in 24 deceased patients with advanced PSCC.

DETAILED DESCRIPTION:
This study focuses on penile squamous cell carcinoma (PSCC), a rare cancer that is more prevalent in underdeveloped regions such as Africa, Asia, and South America, with Brazil having one of the highest incidence rates due to socioeconomic factors. PSCC is primarily associated with risk factors like poor local hygiene, smoking history, phimosis, and human papillomavirus (HPV) infection. The research aims to understand the genomic profiles of PSCC and their correlation with clinical characteristics, particularly in circumcised vs. non-circumcised populations in Brazil. The study will employ next-generation sequencing (NGS) on tumor specimens from 23 deceased patients with advanced PSCC who received treatment in Brazilian cancer sites.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years of age;
* Diagnosis of locally advanced or metastatic squamous-cell penile carcinoma;
* Have received at least one treatment for advanced disease (surgery, radiotherapy and/or chemotherapy);
* Available representative tumor block of formalin-fixed and paraffin-embedded (FFPE) archive, from primary or metastasis;
* Patients must be already deceased at time of data collection.

Exclusion Criteria:

* Patients without medical record available (lost, empty or irretrievable clinical information).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises men aged 18 or older with a diagnosis of locally advanced or metastatic squamous-cell penile carcinoma, who have undergone at least one advanced disease treatment (surgery, radiotherapy, and/or chemotherapy), possess representative tumor blocks from formalin-fixed and paraffin-embedded (FFPE) archives, either from primary or metastatic sites, and are deceased at the time of data collection.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Biomarker Profiling of Penile Carcinoma by NGS | Through study completion, an average of 2 years
  The study employs state-of-the-art molecular analysis methods, including next-generation sequencing (NGS) using a targeted panel (FoundationONE CDx) that assesses 324 genes.

CONTACTS AND LOCATIONS:
Overall Officials: André Poisl Fay, Principal Investigator — PUCRS School of Medicine
Locations (3):
- Brazil (3):
  - Oncocentro Ceará, Fortaleza, Ceará
  - Hospital Universitário da Universidade Federal do Maranhão (UFMA), São Luís, Maranhão
  - Centro de Pesquisa em Oncologia do Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul